CLINICAL TRIAL: NCT02100683
Title: Nit-Occlud PDA Post-Approval Study
Status: Completed | Type: Observational
Sponsor: PFM Medical, Inc (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Other Study IDs: TP126
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Patent Ductus Arteriosus (PDA)
Keywords: Occluder
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PDA Coil: Patients age 6 months to 21 years weighing > 5kg with an angiographically confirmed PDA with a minimum diameter of < 4 mm.
  Interventions: Device: PDA Coil

INTERVENTIONS:
Device: PDA Coil — The Nit-Occlud PDA is a permanently implanted prosthesis indicated for percutaneous, transcatheter closure of small to moderate size patent ductus arteriosus with a minimum angiographic diameter < 4 mm.

SUMMARY:
The Nit-Occlud PDA Post-Approval Study is designed to continue to evaluate the safety and effectiveness of the device in the post-approval phase.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically confirmed PDA with minimum diameter < 4 mm.
* Weight is ≥ 5 kg.
* Age 6 months to 21 years.

Exclusion Criteria:

* Cardiac anomalies requiring surgery.
* Known bleeding or coagulation disorder.
* Febrile illness within 7 days of planned procedure.
* Pregnancy.
* Pulmonary hypertension with increased pulmonary vascular resistance (≥ 5 Wood Units).
* Hypersensitivity to contrast medium.
* Known nickel allergy.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients age 6 months to 21 years weighing >/= 5kg with an angiographically confirmed PDA with a minimum diameter of <4 mm.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Rate of Serious Device and/or Procedure Related Adverse Events as a Measure of Safety | 24 months (2 year)
  The primary safety endpoint is to demonstrate the 24-month serious device-related adverse event rate is no worse than the objective-performance criterion (OPC) of 1%.
Rate of Complete PDA Closure as a Measure of Efficacy | 12 months (1 year)
  The primary effectiveness endpoint is to demonstrate the 12-month (1 year) complete closure rate for the device is no worse than the OPC of 85%. The closure of the ductus arteriosus will be assessed by absence of residual flow at 12 months (1 year) by transthoracic echocardiogram with 2-D color flow mapping and pulse wave Doppler (ECHO).

SECONDARY OUTCOMES:
Rate of Device and/or Procedure Related Adverse Events as a Measure of Safety | 24 months (2 year)
  The secondary safety endpoint is to demonstrate that the rate of device-related adverse events reported through 24-months post procedure is no worse than 6% (OPC rate of 3% plus an added 3% margin).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Levi, MD, Principal Investigator — UCLA Pediatric Cardiology
Locations (11):
- United States (11):
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente, Los Angeles, California
  - Children's Hospital of Central California, Madera, California
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proposed standards for clinical evaluation of patent ductus arteriosus occlusion devices. Multiorganization Advisory Panel to FDA for Pediatric Cardiovascular Devices. Catheter Cardiovasc Interv. 2000 Nov;51(3):293-6. No abstract available. PMID 11066109
- [Result] Kobayashi D, Salem MM, Forbes TJ, Gordon BM, Soriano BD, Dimas V, Goldstein BH, Owada C, Javois A, Bass J, Jones TK, Berman DP, Gillespie MJ, Moore JW, Levi DS. Results of the combined U.S. multicenter postapproval study of the Nit-Occlud PDA device for percutaneous closure of patent ductus arteriosus. Catheter Cardiovasc Interv. 2019 Mar 1;93(4):645-651. doi: 10.1002/ccd.27995. Epub 2018 Dec 3. PMID 30511498